CLINICAL TRIAL: NCT06945562
Title: Influence of Collagen Cone on Jumping Gap Management Around Dental Implants
Acronym: implant
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Faculty of Dental Medicine for Girls (Other Government)
Responsible Party: Principal Investigator, Hala Fathy Abd El Fattah, master's degree student at oral medicine, peridontology ,oral diagnosis and oral Radiology Department, faculty of Dental Medicine for Girls ,Al Azhar university, Faculty of Dental Medicine for Girls
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OMPDR-103-2h
Record Dates: First submitted 2025-04-12; First posted 2025-04-25 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Tooth Loss
Keywords: immediate implant; collagen cone; esthatic zone; jumping gap
MeSH Terms: conditions — Tooth Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Immediate Dental Implant Placement only (Active Comparator): The control group will be assigned for the sites that undergo placement of immediate dental implant (N=8) only.
  Interventions: Procedure: Placement of Immediate Dental Implant Only
- Immediate Dental Implant Placement with Collagen Cone (Active Comparator): The test group include those sites enrolled for placement of immediate dental implant (N=8) with application of collagen cone
  Interventions: Device: collagen cone (resorbable material used for socket sealing )

INTERVENTIONS:
Device: collagen cone (resorbable material used for socket sealing ) — The test group include those sites enrolled for placement of immediate dental implant (N=8) with application of collagen cone
  Arms: Immediate Dental Implant Placement with Collagen Cone
Procedure: Placement of Immediate Dental Implant Only — Participants will receive placement of an immediate dental implant without any additional material (N=8).
  Arms: Immediate Dental Implant Placement only

SUMMARY:
The present study will be performed to assess the clinical and radiographic effect of collagen cone for bone growth in immediate implants.

DETAILED DESCRIPTION:
Improve width and length of buccal plate of alveolar bone, bone density around dental implamts in esthetics zone.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 30-50 years.
* Good general health.
* Adequate bone volume at the implant site.
* Non-compromised periodontal status.

Exclusion Criteria:

* Presence of parafunctional habits (e.g., bruxism, clenching, excessive gum chewing, lip or fingernail biting).
* Smokers.
* Patients receiving chemotherapy or radiotherapy.
* Alcohol or drug abuse.
* Pregnancy and lactation.
* Use of drugs that may affect bone metabolism.

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2025-03-01 (Actual); Study Completion 2025-03-01 (Actual)

PRIMARY OUTCOMES:
Clinical Bleeding Index | from 0 to 9 month
  Assessment of peri-implant soft tissue bleeding using the modified bleeding index:
  0 - No bleeding
  1. - Isolated bleeding spots
  2. - Confluent bleeding
  3. - Profuse bleeding unit of Measure: Score (0-3)
Vertical Bone Loss | from 0 to 9 month
  Measurement of marginal vertical bone height loss around dental implants using CBCT imaging Unit of Measure: Millimeters (mm)
Buccal Plate Width | From 0 to 9 months
  Measurement of buccal bone plate width at the implant site using CBCT. Unit of Measure: Millimeters (mm)

CONTACTS AND LOCATIONS:
Overall Officials: Abeer Gawish, professor, Study Director — Al-Azhar University; lobna Abd-El Aziz, Lecturer, Study Director — Al-Azhar University
Locations (1):
- Hala Fathy Abd El-Fattah Azzam, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No